CLINICAL TRIAL: NCT05319002
Title: Randomized Trial on the Effects of a Group EMDR Intervention on Narrative Complexity and Specificity of Autobiographical Memories: a Path Analytic and Supervised Machine Learning Approach
Brief Title: Effects of a Group EMDR Intervention on Narrative Complexity and Specificity of Autobiographical Memories: the Hug the Child Study (HTC)
Acronym: HTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Andrea Poli, Principal Investigator, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HTC-01
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Child, Only; Narration; Memory Dysfunction; Distress, Emotional; Cognitive Change
Keywords: Child; EMDR; Narrative complexity; Autobiographical memories; Distress; Cognition
MeSH Terms: conditions — Narration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EMDR (Experimental): Participants in the experimental group will undergo a 3-week group EMDR intervention with weekly 60-minute group sessions.
  Interventions: Behavioral: Group EMDR
- Control (No Intervention): The control group will follow routine daily school activities

INTERVENTIONS:
Behavioral: Group EMDR — The eight phases of the adapted group EMDR protocol was administered during each session: 1. Meeting: Explaining the nature of trauma, group rules, name tags, filling in the scales. 2. Preparation: Exploring children's support system, explaining EMDR, safe place, resource exercise, and installation with bilateral stimulation (BLS, butterfly hug or knee tapping). 3. Assessment: Drawing the worst image on a small separate sheet of paper, SUD level, (negative cognition, emotions, body sensations - if possible). 4. Desensitization: It is done with drawing on 4 separate papers with BLS (butterfly hug or knee tapping). 5. Installation: With the healing story written according to the adaptive information processing (AIP) model, the installation is accompanied BLS. 6. Body scan: A positive body state is installed with the relaxation technique. 7. Closure & future template: Strong closure with artwork. 8. Re-evaluation: if possible.
  Arms: Group EMDR

SUMMARY:
Background and study aims:

The Eye Movement Desensitization and Reprocessing Group Protocol with Children (EMDR-GP/C) was first developed by Korkmazlar following the Marmara earthquake in Turkey in 1999 and can be adapted for different populations. The aim of this study is to assess if a EMDR-GP program may help primary school students in improving narrative complexity and specificity of autobiographical memories, as well as their subjective unit of distress (SUD) and validity of cognition (VoC).

Who can participate? Students attending the fourth or fifth year of primary school

What does the study involve? Participants will be randomly assigned to the experimental and control groups. Participants in the experimental group will undergo a 3-week EMDR-GP with weekly 60-minute group sessions (3 sessions), while the control group will follow routine daily school activities.

Questionnaires will be used to assess narrative complexity, specificity of autobiographical memories, SUD and VoC before and after the intervention.

What are the possible benefits and risks of participating? Benefits of participating in the study may include an improvement of narrative complexity, specificity of autobiographical memories, and their SUD and VoC.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 9 to 11 years
2. Children have reasonable comprehension of spoken language and can follow simple instructions
3. Children and their parents are willing to attend all intervention sessions
4. Children and parents have an adequate understanding of Italian

Exclusion Criteria:

1. Concurrent enrollment in other intervention trials
2. Child regularly practices EMDR intervention, or other therapeutical interventions, such as cognitive behavioral therapy or meditation.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Event coding - Pre-intervention | Event coding is measured before the 3-week group EMDR intervention
  Event coding is measured using Manual for Coding Events in Self Defining Memories. "Relationship" nominal score means a better outcome
Memory specificity level - Pre-intervention | Memory specificity level is measured before the 3-week group EMDR intervention
  Memory specificity level is measured using Classification System and Scoring for Self-defining Autobiographical Memories. "Specific" nominal score means a better outcome
Narrative complexity level - Pre-intervention | Narrative complexity level is measured before the 3-week group EMDR intervention
  Narrative complexity level is measured using Coding System for autobiographical Memory Narratives in Psychotherapy. Higher scores mean a better outcome.
Subjective Unit of Distress - Pre-intervention | Subjective Unit of Distress is measured before the 3-week group EMDR intervention
  Subjective Unit of Distress is measured using a self-reporting scale with a 0- to 10-point rating scale. Higher scores mean a worse outcome
Validity of Cognition - Pre-intervention | Validity of Cognition is measured before the 3-week group EMDR intervention
  Validity of Cognition is measured using a self-reporting scale with a 1- to 7-point rating scale. Higher scores mean a better outcome
Event coding - Post-intervention | Event coding is measured after the 3-week group EMDR intervention
  Event coding is measured using Manual for Coding Events in Self Defining Memories. "Relationship" nominal score means a better outcome
Memory specificity level - Post-intervention | Memory specificity level is measured after the 3-week group EMDR intervention
  Memory specificity level is measured using Classification System and Scoring for Self-defining Autobiographical Memories. "Specific" nominal score means a better outcome
Narrative complexity level - Post-intervention | Narrative complexity level is measured after the 3-week group EMDR intervention
  Narrative complexity level is measured using Coding System for autobiographical Memory Narratives in Psychotherapy. Higher scores mean a better outcome.
Subjective Unit of Distress - Post-intervention | Subjective Unit of Distress is measured after the 3-week group EMDR intervention
  Subjective Unit of Distress is measured using a self-reporting scale with a 0- to 10-point rating scale. Higher scores mean a worse outcome
Validity of Cognition - Post-intervention | Validity of Cognition is measured after the 3-week group EMDR intervention
  Validity of Cognition is measured using a self-reporting scale with a 1- to 7-point rating scale. Higher scores mean a better outcome

SECONDARY OUTCOMES:
Autobiographical memory definition - Pre-intervention | Autobiographical memory definition is measured before the 3-week group EMDR intervention
  Autobiographical memory definition is measured using Coding System for Autobiographical Memory Narratives in Psychotherapy. "Autobiographic" nominal score means a better outcome.
Memory integration level - Pre-intervention | Memory integration level is measured before the 3-week group EMDR intervention
  Memory integration level is measured using Classification System and Scoring for Self-defining Autobiographical Memories. "Integrated" nominal score means a better outcome
Autobiographical memory definition - Post-intervention | Autobiographical memory definition is measured after the 3-week group EMDR intervention
  Autobiographical memory definition is measured using Coding System for Autobiographical Memory Narratives in Psychotherapy. "Autobiographic" nominal score means a better outcome.
Memory integration level - Post-intervention | Memory integration level is measured after the 3-week group EMDR intervention
  Memory integration level is measured using Classification System and Scoring for Self-defining Autobiographical Memories. "Integrated" nominal score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Poli, Psy.D., Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
Raw data are available on request.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Poli A, Gemignani A, Miccoli M. Randomized Trial on the Effects of a Group EMDR Intervention on Narrative Complexity and Specificity of Autobiographical Memories: A Path Analytic and Supervised Machine-Learning Study. Int J Environ Res Public Health. 2022 Jun 23;19(13):7684. doi: 10.3390/ijerph19137684. PMID 35805348